CLINICAL TRIAL: NCT00798148
Title: Evaluation of Benefit and Side Effects of 131I-MIBG in Combination With Myeloablative Chemotherapy and Autologous Peripheral Blood Stem Cell Transplantation for the Treatment of High-risk Neuroblastoma
Brief Title: 131I-MIBG With Myeloablative Chemotherapy and Autologous Stem Cell Transplantation for the Treatment of High-risk Neuroblastoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87-01-36-6853
Record Dates: First submitted 2008-11-23; First posted 2008-11-25 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; MIBG; Autologous Peripheral Stem Cell Transplantation
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; Etoposide; Melphalan; Carboplatin

ARMS (1):
- MIBG (Experimental)
  Interventions: Drug: 131I-MIBG , Etoposide, Melphalan, Carboplatin, Autologous Peripheral Stem Cell Transplantation

INTERVENTIONS:
Drug: 131I-MIBG , Etoposide, Melphalan, Carboplatin, Autologous Peripheral Stem Cell Transplantation — 131I-MIBG 12mci/kg CEM(Etoposide)=1200mg/m2 Melphalan=210mg/m2 Carboplatin=1500mg/m2 Autologous Peripheral Stem Cell Transplantation

SUMMARY:
This trial is studying how well iodine I 131 metaiodobenzylguanidine together with combination chemotherapy works in treating patients who are undergoing an autologous peripheral stem cell for high risk or relapsed neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Neuroblastoma and/or demonstration of tumor cells in bone marrow with elevated urinary catecholamine metabolites
* High risk according COG (Children Oncology Group)OR Relapse OR Refractory
* As at least one I131-MIBG avid target lesion determined by diagnostic MIBG scan
* Glomerular filtration rate or creatinine clearance > 60 ml/min
* No tumor cell in Bone Marrow by routine morphology aspiration and biopsy before peripheral stem cell collection
* No active infection

Exclusion Criteria:

* Impaired renal function
* No avid I131-MIBG lesion
* Active infection

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Response (complete response, very good partial response, and partial response) at one-years post stem cell transplantation | one-years post stem cell transplantation

SECONDARY OUTCOMES:
Overall survival | one-year after stem cell tranplantation

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Hematology-Oncology & SCT Research Center, Tehran, Tehran Province
  - Research Institute for Nuclear Medicine, Tehran, Tehran Province